CLINICAL TRIAL: NCT00003483
Title: Phase II Study of Antineoplastons A10 and AS2-1 in Patients With Meningioma
Brief Title: Antineoplaston Therapy in Treating Patients With Meningioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Burzynski Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066521; BC-BT-28 (Other: Burzynski Research Institute, Inc.)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2017-02-17 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-07

CONDITIONS: Meningioma
Keywords: adult meningioma; recurrent adult meningioma
MeSH Terms: conditions — Meningioma | interventions — antineoplaston A10; antineoplaston AS 2-1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antineoplaston therapy (Experimental): Antineoplaston therapy (Atengenal + Astugenal) by IV infusion every four hours for at least 12 months. Study subjects receive increasing dosages of Atengenal and Astugenal until the maximum tolerated dose is reached.
  Interventions: Drug: Antineoplaston therapy (Atengenal + Astugenal)

INTERVENTIONS:
Drug: Antineoplaston therapy (Atengenal + Astugenal) — Adults with a meningioma will receive Antineoplaston therapy (Atengenal + Astugenal).
  Other Names: A10 (Atengenal); AS2-1 (Astugenal)

SUMMARY:
RATIONALE: Current therapies for adults with meningioma provide limited benefit to the patient. The anti-cancer properties of Antineoplaston therapy suggest that it may prove beneficial in the treatment of adults with meningioma.

PURPOSE: This study is being performed to determine the effects (good and bad) that Antineoplaston therapy has on adults with meningioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the efficacy of Antineoplaston therapy in adults with meningima as measured by an objective response to therapy (complete response, partial response) or stable disease.
* To determine the safety and tolerance of Antineoplaston therapy in adults with meningima.

OVERVIEW: This is a single arm, open-label study in which adults with meningioma receive gradually escalating doses of intravenous Antineoplaston therapy (Atengenal + Astugenal) until the maximum tolerated dose is reached. Treatment continues for at least 12 months in the absence of disease progression or unacceptable toxicity. After 12 months, patients with a complete or partial response or with stable disease may continue treatment.

To determine objective response, tumor size is measured utilizing MRI scans, which are performed every 8 weeks for the first two years, every 3 months for the third and fourth years, every 6 months for the 5th and sixth years, and annually thereafter.

PROJECTED ACCRUAL: A total of 20-40 patients will be accrued to this study

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed meningioma that has progressed or recurred following surgical resection and radiotherapy
* Evidence of residual tumor by MRI scan performed within two weeks prior to study entry

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* At least 2 months

Hematopoietic:

* Hemoglobin at least 9 g/dL
* WBC at least 2000/mm3
* Platelet count at least 50,000/mm3

Hepatic:

* Bilirubin no greater than 2.5 mg/dL
* SGOT/SGPT no greater than 5 times upper limit of normal
* No hepatic failure

Renal:

* Creatinine no greater than 2.5 mg/dL
* No history of renal conditions that contraindicate high dosages of sodium

Cardiovascular:

* No chronic heart failure
* No uncontrolled hypertension
* No history of congestive heart failure
* No history of other cardiovascular conditions that contraindicate high dosages of sodium

Pulmonary:

* No serious lung disease, such as chronic obstructive pulmonary disease

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 4 weeks after study
* No active infection
* No other serious concurrent disease

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy and recovered
* No concurrent immunomodulatory agents

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No concurrent antineoplastic agents

Endocrine therapy:

* Concurrent corticosteroids allowed
* At least 4 weeks since prior therapy with mifepristone and recovered

Radiotherapy:

* At least 8 weeks since prior radiotherapy and recovered

Surgery:

* Recovered from prior surgery

Other:

* Prior cytodifferentiating agent allowed
* No prior antineoplaston therapy

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 1998-06; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanislaw R. Burzynski, MD, PhD, Principal Investigator — Burzynski Research Institute
Locations (1):
- Burzynski Clinic, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Burzynski Research Institute — http://www.burzynskiresearch.com
- See also: Burzynski Clinic — http://www.burzynskiclinic.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three patients were recruited between June 1996 and March 2004. All study subjects were seen at the Burzynski Clinic in Houston TX
Period: Overall Study
Arm/Group | Antineoplaston Therapy
Started | 3
Completed | 2
Not Completed | 1
Not completed — Not evaluable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 3
Age, Continuous [Median (Full Range); unit: Years] | 41.8 [30.2 to 49.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response
Description: Objective response rate per Response Assessment in Neuro-Oncology (RANO) for target lesions and assessed by MRI: Complete Response (CR), disappearance of all disease sustained for at least four weeks; Partial Response (PR), >=50% decrease in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least four weeks; Stable Disease (SD), <50% decrease and <25% increase in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions, sustained for at least eight weeks; Progressive Disease (PD), >=25% increase in the sum of the products of of the greatest perpendicular diameters of all measurable enhancing lesions.
Time Frame: 12 months
Measure: Number; unit: Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 2
Participants
  Stable Disease | 2
  Objective Response | 0

2. Secondary Outcome: Percentage of Participants Who Survived
Description: 6 months, 12 months, 24 months overall survival
Time Frame: 6 months, 12 months, 24 months
Population: All study subjects receiving any Antineoplaston therapy
Measure: Number; unit: Percentage of Participants
Arm/Group | Antineoplaston Therapy
Number analyzed (Participants) | 3
Percentage of Participants
  6 months overall survival | 66.7
  12 months overall survival | 33.3
  24 months overall survival | 33.3

ADVERSE EVENTS:
Time Frame: 7 years, 9 months
Description: Three patients were recruited between June 1996 and March 2004. All study subjects were seen at the Burzynski Clinic in Houston TX
Arm/Group | Antineoplaston Therapy
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=3)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 1 — The Allergic reaction/hypersensitivity (including drug fever) was possibly related to Antineoplaston therapy.
Infection (documented clinically): Skin (cellulitis) (Infections and infestations) | 1 — The Infection (documented clinically): Skin (cellulitis) was not related to Antineoplaston therapy.
Confusion (Nervous system disorders) | 1 — The Confusion was not related to Antineoplaston therapy.
Somnolence/depressed level of consciousness (Nervous system disorders) | 1 — The Somnolence/depressed level of consciousness was not related to Antineoplaston therapy.
Pain: Head/headache (Nervous system disorders) | 1 — The Pain: Head/headache was not related to Antineoplaston therapy.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Antineoplaston Therapy (N=3)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 2
Lymphopenia (Blood and lymphatic system disorders) | 1
Central Venous Catheter Infection (Infections and infestations) | 2
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2
Weight gain (General disorders) | 1
Edema/Fluid retention (General disorders) | 1
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 1
Infection (documented clinically): Mucosa (Infections and infestations) | 1
Infection (documented clinically): Skin (cellulitis) (Infections and infestations) | 1
Infection (documented clinically): Upper airway NOS (Infections and infestations) | 1
Opportunistic infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No